CLINICAL TRIAL: NCT06805110
Title: Improving the Accuracy of Malaria RDT Reporting in Public Primary Healthcare Facilities in Nigeria
Brief Title: MaCRA Part B in Nigeria
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: USAID termination of project funding and activities
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Sydani Group (Unknown); US President's Malaria Initiative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RES-00850
Record Dates: First submitted 2025-01-22; First posted 2025-02-03 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monthly RDT validation during DHIS2 data review meetings (Experimental): The Nigeria national malaria program will lead monthly RDT validation at selected legal government areas (LGAs). Health facilities will be asked to retain all RDT cassettes performed for the prior month and bring them to a monthly validation meeting. During these meetings, RDT cassettes will be scanned using the HealthPulse application, which will automatically tally the number of RDTs by brand and result. The application will also allow for the entry of aggregated testing data, including the total number of tests conducted and the RDT results recorded in the health facility register. Discrepancies between the HealthPulse data and facility records will be calculated, with a focus on identifying and addressing discrepancies exceeding a designated threshold (e.g., 10%) that takes into account the proportion of cassettes that may have changed results over the past month. Facilities with significant discrepancies may undergo a detailed audit to align RDT cassettes with patient records.
  Interventions: Behavioral: Monthly RDT validation during DHIS2 data review meetings
- Control (No Intervention): There will be no new activities in the control facilities.

INTERVENTIONS:
Behavioral: Monthly RDT validation during DHIS2 data review meetings — The Nigeria national malaria program will lead monthly RDT validation at selected legal government areas (LGAs). Health facilities will be asked to retain all RDT cassettes performed for the prior month and bring them to a monthly validation meeting. During these meetings, RDT cassettes will be scanned using the HealthPulse application, which will automatically tally the number of RDTs by brand and result. The application will also allow for the entry of aggregated testing data, including the total number of tests conducted and the RDT results recorded in the health facility register. Discrepancies between the HealthPulse data and facility records will be calculated, with a focus on identifying and addressing discrepancies exceeding a designated threshold (e.g., 10%) that takes into account the proportion of cassettes that may have changed results over the past month. Facilities with significant discrepancies may undergo a detailed audit to align RDT cassettes with patient records.
  Arms: Monthly RDT validation during DHIS2 data review meetings

SUMMARY:
This study aims to evaluate the effectiveness of monthly malaria rapid diagnostic test (RDT) validation meetings at district level on reducing the proportion of RDT results recorded as positive in health facility registers in Nigeria.

DETAILED DESCRIPTION:
PMI Insights supported a multi-country evaluation of the accuracy of the recording and reporting of rapid diagnostic test (RDT) results at health facilities in Benin, Côte d'Ivoire, Nigeria, and Uganda (MaCRA Part A). The evaluation found a high degree of agreement between RDT results recorded in health facilities and an objective panel reading of the same RDTs. However, the changes in test positivity rate (TPR) after the start of the study suggest that some of this agreement may have been a result of the Hawthorne effect: in all countries except Benin, TPR declined after the start of the evaluation in facilities where evaluation staff were present, compared with control facilities. This suggests that the presence of evaluation staff caused health care workers to change their behavior with respect to reporting positive RDT results. The study evaluated the durability of RDT results and found that 95% of RDT cassettes retained their original reading over a one-month period. This provides evidence that stored RDT cassettes may be compared to health facility registers at monthly validation meetings, as long as a certain margin of error is used to account for the proportion of tests that may change.

The results from the first phase of the study were used to identify potential interventions to improve RDT reporting and recording accuracy in health facilities. The second phase of the study aims to evaluate the effectiveness of monthly district-level RDT result validation meetings on reducing the proportion of RDT results recorded as positive in health facility registers and reported to the national health management information system.

This is a two-arm cluster-randomized controlled effectiveness evaluation. Districts will serve as the clusters and will be assigned using restricted randomization to the intervention or control arm. In the intervention arm, the Ministry of Health will lead monthly district-level RDT validation meetings facilitated by a digital phone-based app which uses AI to record RDT results (HealthPulse, Audere, Johannesburg, South Africa). There will be no study activities in the control facilities.

Monthly RDT validation meetings will take place over a four-month period (April to July 2025), after which a cross-sectional survey and in- depth interviews will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers responsible for testing or interpreting malaria RDTs in the selected study facilities
* LGA health teams involved in the monthly RDT validation meetings from LGAs selected for the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of RDT results reported as positive from study facilities on the DHIS2 | 4 months (April - July 2025)
  Data for the intervention and control facilities will be downloaded from the DHIS2 at the end of August 2025

SECONDARY OUTCOMES:
Ratio of TPR between health facility registers and RDT cassettes in intervention facilities over time. | 4 months (April - July 2025)
  The change in ratio will be measured by using the TPR from the facility registers and the TPR from the cassettes entered into the HealthPulse app
Total costs associated with monthly RDT validation exercises | 4 months (April - July 2025)
  Collection and analysis of cost data, including personnel costs, travel expenses, and other project-related expenses will be used to estimate the total costs associated with the validation meetings
HCWs subjective norms, attitudes, perceptions and practices regarding RDT usage | Immediately after intervention period (August 2025)
  A questionnaire will be administered to HCWs in the intervention and control group to compare differences in their subjective norms, attitudes, perceptions and practices regarding RDT
Acceptability and feasibility of implementing monthly RDT validation exercises | Immediately after intervention period (August 2025)
  In-depth interviews will be conducted with HCWs, local government areas (LGAs) and state officials to understand their perceptions of the acceptability of the monthly validation processes
Acceptability and feasibility of using a digital smartphone application for monthly RDT validation exercises | Immediately after intervention period (August 2025)
  In-depth interviews will be conducted with HCWs, LGA and state officials to understand their perceptions of the acceptability and feasibility of using the digital application during monthly validation

CONTACTS AND LOCATIONS:
Overall Officials: Sunday Atobatele, Principal Investigator — Sydani Group